CLINICAL TRIAL: NCT00123825
Title: A Phase II Trial of Gemcitabine and Cisplatin In Unresectable Or Metastatic Biliary Tract and Gallbladder Cancer
Brief Title: Gemcitabine and Cisplatin for Gallbladder and Biliary Tract Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other); Massachusetts General Hospital (Other); Beth Israel Deaconess Medical Center (Other); Eli Lilly and Company (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 02-065
Record Dates: First submitted 2005-07-25; First posted 2005-07-26 (Estimated); Last update posted 2007-12-21 (Estimated); Status verified 2007-12

CONDITIONS: Gallbladder Cancer; Biliary Tract Cancer
Keywords: Gallbladder; Biliary Tract; Cholangiocarcinoma
MeSH Terms: conditions — Gallbladder Neoplasms; Biliary Tract Neoplasms; Cholangiocarcinoma | interventions — Gemcitabine; Cisplatin

INTERVENTIONS:
Drug: Gemcitabine
Drug: Cisplatin

SUMMARY:
In the United States, the incidence of biliary tract cancer and gallbladder cancer has been estimated to be 6,000-8,000 patients per year. Currently, there is no standard therapy for these tumors once the disease has spread and is inoperable. Recent small studies with gemcitabine have shown a positive response rate. The investigators plan to test the combination of gemcitabine with cisplatin for biliary tract and gallbladder cancers.

DETAILED DESCRIPTION:
Gemcitabine and cisplatin will be administered weekly for two weeks (on day 1 and day 8) followed by a one week rest period (1 cycle is 3 weeks). On day one and eight of each cycle the patient will have a physical exam and blood work. During the first two cycles, additional blood work will be drawn on day 15 as well. Reassessment of the tumor will be performed at 6 weeks, 12 weeks, and every 9 weeks thereafter. Patients will remain on treatment until further evidence of disease progression or unacceptable side effects occur.

ELIGIBILITY:
Inclusion Criteria:

* Histologically-confirmed, locally unresectable or metastatic biliary tract (bile ducts, hepatic duct, cystic duct, common bile duct, ampulla of Vater) or gallbladder adenocarcinoma. Patients must have at least one measurable lesion greater than 1 cm, by Response Evaluation Criteria in Solid Tumors (RECIST) criteria outside of prior radiation field.
* Zero to one prior chemotherapy for biliary tract or gallbladder cancer. Prior chemoembolization to the liver allowed as long as measurable disease is outside of chemoembolization area and other baseline characteristics are met. No prior gemcitabine or cisplatin therapy allowed.
* No chemotherapy within past 3 weeks of initiation of therapy (6 weeks if prior therapy was mitomycin C or nitrosurea)
* Chronological age > 18 years.
* ECOG performance status 0-2; life expectancy >12 weeks.
* Laboratory values: ANC greater than or equal to 1500/mm3; platelets greater than or equal to 100,000/mm3; SGOT and SGPT less than or equal to 3x upper limits of normal (unless liver is involved with tumor, in which case the transaminases must be less than or equal to 5 x upper limits of normal); total bilirubin less than or equal to 2.0 mg/dL.
* Creatinine less than or equal to 1.8 mg/dL or creatinine clearance greater than or equal to 50 mL/min
* All patients must sign informed consent.
* Patients may have prior placement of stents or shunts to relieve obstruction.

Exclusion Criteria:

* Patients with either clinically apparent central nervous system metastases or carcinomatous meningitis.
* Myocardial infarction in the past six months.
* Major surgery in the past two weeks.
* Uncontrolled serious medical or psychiatric illness.
* Women must not be pregnant or lactating. Both men and women of childbearing potential must be advised of the importance of using effective birth control measures during the course of the study.
* Patients with concurrent malignancy of any site, except for limited basal cell carcinoma or squamous cell carcinoma of the skin or carcinoma in situ of the cervix; patients with any other malignancy within 5 years of study entry, except for curatively treated basal cell carcinoma or squamous cell carcinoma of the skin or carcinoma in situ of the cervix.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2002-07; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
To determine the response rate of the combination gemcitabine and cisplatin in patients with advanced biliary tract and gallbladder cancers

SECONDARY OUTCOMES:
To determine the overall survival rate, progression-free survival rate, time to progression and duration of response
To determine the toxicity of gemcitabine and cisplatin
To assess the biomarker CA 19-9 response to the regimen and to correlate the CA 19-9 response with radiologic response and survival

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey A Meyerhardt, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts